CLINICAL TRIAL: NCT04298840
Title: Influence of Creatine Monohydrate Supplementation on Androgens and Global Hair Assessments
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor indicated it was unable/unwilling to support project at the present time.
Sponsor: Texas Tech University (Other)
Collaborators: Legion Athletics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2019-997
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Dihydrotestosterone; Testosterone; Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive creatine monohydrate or placebo for daily consumption during the study period.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Monohydrate (Experimental)
  Interventions: Dietary Supplement: Creatine Monohydrate Supplementation
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Supplementation

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate Supplementation — Participants in the creatine monohydrate supplementation arm will consume 5 grams per day of creatine monohydrate.
  Arms: Creatine Monohydrate
Dietary Supplement: Placebo Supplementation — Participants in the placebo supplementation arm will consume 5 grams per day of maltodextrin placebo.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial examining the effects of creatine monohydrate supplementation on androgens and hair loss in free-living adult males. Participants will complete 6 months of supplementation of 5 grams per day of creatine monohydrate while following their normal lifestyle practices. At baseline and six months after study initiation, participants will complete laboratory assessments. These assessments will include a standard blood draw for evaluation of total testosterone (T), free T, dihydrotestosterone (DHT), and DHT:T ratios in the blood, as well as global photography and questionnaires to evaluate hair loss. This study will examine the claim that creatine increases DHT concentrations and and DHT:T ratio, as well as provide novel data regarding whether creatine promotes hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Male between the ages of 18 and 35
* Weight of at least 110 pounds
* Generally healthy (defined as an absence of a disease or medical condition which could potentially be negatively influenced by study participation or confound study results)
* Low levels of habitual creatine consumption, defined as consuming an average of <10 g/week of creatine from all supplemental sources within the three months prior to study initiation
* Willingness to report to baseline and final assessments with a similar haircut (i.e. willingness to replicate baseline haircut prior final assessment, to the best of his ability) and one that allows for evaluation of hair growth patterns (e.g., not a completely shaved head that disallows visualization of the hairline)
* Willingness to adhere to the supplementation protocol for the duration of the study (i.e., 6 months of daily supplementation with 5 grams per day of creatine monohydrate or placebo) and abstain from additional creatine supplement ingestion during this time.
* Willingness to abstain from any treatments related to hair loss or hair growth for the duration of the study
* Willingness to maintain normal practices regarding hair products (i.e. continue to use regular shampoo, conditioner, and other products over the duration of the study and abstain from switching products during the study if at all possible)

Exclusion Criteria:

* Failing to meet any of the aforementioned inclusion criteria
* Presence of pacemaker or any electrical device (due to electrical currents administered by bioimpedance devices used to assess body composition)
* Individual currently participates in any type of hair loss treatment or procedure or has undergone any such treatment or procedure within the last 12 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Dihydrotestosterone | 6 months
  Blood concentration of dihydrotestosterone.
Dihydrotestosterone-to-Testosterone Ratio 1 | 6 months
  Ratio of dihydrotestosterone to total testosterone in the blood.
Dihydrotestosterone-to-Testosterone Ratio 2 | 6 months
  Ratio of dihydrotestosterone to free testosterone in the blood.
Total Testosterone | 6 months
  Total testosterone in the blood.
Free Testosterone | 6 months
  Free testosterone in the blood.
Global Hair Assessments | 6 months
  Subjectively scored assessment of changes in hair properties from baseline to the end of the intervention. Assessor will be a blinded expert.

SECONDARY OUTCOMES:
Self-Reported Hair Assessments | 6 months
  Survey allowing for participant-reported changes in hair properties as a result of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Grant M Tinsley, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Department of Kinesiology & Sport Management, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Merwe J, Brooks NE, Myburgh KH. Three weeks of creatine monohydrate supplementation affects dihydrotestosterone to testosterone ratio in college-aged rugby players. Clin J Sport Med. 2009 Sep;19(5):399-404. doi: 10.1097/JSM.0b013e3181b8b52f. PMID 19741313
- [Background] Kreider RB, Kalman DS, Antonio J, Ziegenfuss TN, Wildman R, Collins R, Candow DG, Kleiner SM, Almada AL, Lopez HL. International Society of Sports Nutrition position stand: safety and efficacy of creatine supplementation in exercise, sport, and medicine. J Int Soc Sports Nutr. 2017 Jun 13;14:18. doi: 10.1186/s12970-017-0173-z. eCollection 2017. PMID 28615996
- [Background] Kaufman KD. Androgens and alopecia. Mol Cell Endocrinol. 2002 Dec 30;198(1-2):89-95. doi: 10.1016/s0303-7207(02)00372-6. PMID 12573818
- [Background] Trueb RM. Molecular mechanisms of androgenetic alopecia. Exp Gerontol. 2002 Aug-Sep;37(8-9):981-90. doi: 10.1016/s0531-5565(02)00093-1. PMID 12213548
- [Background] Bang HJ, Yang YJ, Lho DS, Lee WY, Sim WY, Chung BC. Comparative studies on level of androgens in hair and plasma with premature male-pattern baldness. J Dermatol Sci. 2004 Feb;34(1):11-6. doi: 10.1016/j.jdermsci.2003.11.005. PMID 14757277
- [Background] Olsen EA, Whiting DA, Savin R, Rodgers A, Johnson-Levonas AO, Round E, Rotonda J, Kaufman KD; Male Pattern Hair Loss Study Group. Global photographic assessment of men aged 18 to 60 years with male pattern hair loss receiving finasteride 1 mg or placebo. J Am Acad Dermatol. 2012 Sep;67(3):379-86. doi: 10.1016/j.jaad.2011.10.027. Epub 2012 Feb 9. PMID 22325459
- [Background] Van Neste MD. Assessment of hair loss: clinical relevance of hair growth evaluation methods. Clin Exp Dermatol. 2002 Jul;27(5):358-65. doi: 10.1046/j.1365-2230.2002.01003.x. PMID 12190635
- [Background] Ashique K, Kaliyadan F. Clinical photography for trichology practice: tips and tricks. Int J Trichology. 2011 Jan;3(1):7-13. doi: 10.4103/0974-7753.82118. PMID 21769229
- [Background] Norwood OT. Male pattern baldness: classification and incidence. South Med J. 1975 Nov;68(11):1359-65. doi: 10.1097/00007611-197511000-00009. PMID 1188424
- [Background] Gupta M, Mysore V. Classifications of Patterned Hair Loss: A Review. J Cutan Aesthet Surg. 2016 Jan-Mar;9(1):3-12. doi: 10.4103/0974-2077.178536. PMID 27081243